CLINICAL TRIAL: NCT07107984
Title: Assessment of Physical Performance in Obese, Overweight, and Normal-Weight Children
Brief Title: Assessment of Physical Performance in Children
Status: Active, not recruiting | Type: Observational
Sponsor: Afyonkarahisar Health Sciences University (Other)
Responsible Party: Principal Investigator, Gülşen Taşkın, Assistant Professor, Afyonkarahisar Health Sciences University
Other Study IDs: 2025/8
Record Dates: First submitted 2025-07-24; First posted 2025-08-06 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Physical Performance

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Overweight children: Same researcher will carry the same evaluation procedures for overweight and normal-weight children registered at the Sports Center. Demographic and anthropometric characteristics such as age, sex, height, weight, waist circumference, and hip circumference will be measured mass index (BMI) and waist-to-hip ratio will be calculated. Scores from the one-leg balance test, agility test, standing long jump test, and 30-second sit-to-stand test will also be collected. In the study, only the initial measurements of children who applied to the Sports Center will be used.
- Obese Children: In the first stage of the study, data on age, sex, height, weight, waist circumference, and hip circumference of obese children will be collected from the archives of the Physiotherapy Services Unit at the Healthy Life Center (HLC).Body mass index (BMI) and waist-to-hip ratio will be calculated. Scores from the one-leg balance test, agility test, standing long jump test, and 30-second sit-to-stand test will also be collected. Entire data of obese children will be retrieved from the unit's archives. No new assessments will be conducted.
- Normal-Weight Children: Same researcher will carry the same evaluation procedures for overweight and normal-weight children registered at the Sports Center. Demographic and anthropometric characteristics such as age, sex, height, weight, waist circumference, and hip circumference will be measured mass index (BMI) and waist-to-hip ratio will be calculated. Scores from the one-leg balance test, agility test, standing long jump test, and 30-second sit-to-stand test will also be collected. In the study, only the initial measurements of children who applied to the Sports Center will be used.

SUMMARY:
Overweight and obesity are defined as abnormal or excessive fat buildup that may affect health . Body mass index(BMI) is the main property to define and classify the obesity . One of the most considerable public health problem of the 21st century is childhood obesity . Based on the worldwide estimation in 2016, 124 million children and adolescents aged between 5 and 19 were obese, and there were 213 million overweight individuals.

The health complications associated with overweight and obesity in childhood-often not noticeable until adulthood-include cardiovascular diseases (particularly heart disease and stroke), diabetes, musculoskeletal disorders (especially osteoarthritis), and certain types of cancer (endometrial, breast, and colon). Engaging in screen time of more than 2-3 hours per day reduces physical activity levels and increases food intake in children. A study in Turkey reported that 36.2% of children aged between 6 to 9, spend more than two hours per day watching TV or using a computer on weekdays, and this rate increases to 69.9% on weekends. There are revised regional reference values accessible for the anthropometric assessment of Turkish children. Health-related physical fitness in children is correlated with flexibility, muscular and cardiovascular endurance, muscular strength, and body composition. Also, performance-related or sport-specific abilities are associated to agility, power, speed, coordination, and balance. Sevimay implemented the motor performance test (agility parameter) in 1986, which is developed by Morris, Atwater, Williams and Wilmore in 1980, on 205 children aged between 3 and 6. In this study, same test is applied to assess motor performance in children. In order to assess static balance with minimal equipment, the One-leg standing test is used. To assess lower extremity motor performance, the 30-Second Sit-to-Stand Test was used . Evaluation of physical performance levels of obese, overweight, and normal-weight children is the aim of this study.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 6 and 11 years
* Informed consent provided by their parents

Exclusion Criteria:

* Children with orthopedic, neurological, psychological or cognitive disorders
* Children whose parents do not consent to participation or later withdraw their consent

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: This descriptive research will be organized with primary school students aged 6 to 11
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-07-10 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The one-leg stance test. | baseline
  Balance will be evaluated using the one-leg stance test. The test result will be recorded as standing time on one leg (seconds).
Agility | Baseline
  Agility will be evaluated using agility the test. The test result will be recorded in seconds.
The standing long jump test | Baseline
  Muscular strength will be evaluated with the standing long jump. The test result will be recorded in centimeters.
The 30-second sit-to-stand test | Baseline
  Lower extremity motor performance will be evaluated using the 30-second sit-to-stand test. At the end of the test, the number of times they sit and stand for 30 seconds will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Afyonkarahisar Health Science University, Afyonkarahisar, Afyonkarahisar, Turkey (Türkiye)